CLINICAL TRIAL: NCT00883376
Title: Classification of Stanford for Snore as Factor of Aggravation of the AIH in Patients With OSAS.
Brief Title: Classification of Stanford for Snore as Factor of Aggravation of the Apnea Hypopnea Index (AIH) in Patients With Obstructive Sleep Apnea Syndrome (OSAS)
Acronym: StanforAIH
Status: Completed | Type: Observational
Sponsor: Irmandade da Santa Casa de Misericoridia de Limeira (Other)
Responsible Party: Marcos Marques Rodrigues, Irmandade da Santa Casa de Misericoridia de Limeira
Other Study IDs: CEP ISCML 114/08; StanforAIH
Record Dates: First submitted 2009-04-16; First posted 2009-04-17 (Estimated); Last update posted 2009-04-17 (Estimated); Status verified 2009-04

CONDITIONS: Obstructive Sleep Apnea Syndrome
Keywords: Classification of Stanford for Snoring; OSAS; Apnea-Hipopnea Index
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: OSAS patients
- 2: no OSAS patients

SUMMARY:
Introduction: Obstructive sleep apnea syndrome (OSAS) became an important and prevalent illness in recent years. The population occidental becomes fat each time, and this symptom is associated the biggest risk for the OSAS. Snore presence is extremely associated with OSAS. Snoring is present in about 90 - 95% of the patients with OSAS.

Objectives: Evaluate the influence in the Stanford classification as predictor factor of gravity of the OSAS.

Materials and Methods: They evaluated and classified 107 patients, Classification of Mallampati, Friedman, Classification of Stanford and how much the gravity of the OSAS for the AIH.

ELIGIBILITY:
Inclusion Criteria:

* Not exhibiting any exclusion criteria
* Age > 21 years

Exclusion Criteria:

* Nasal tumor
* BMI >40
* Nasal polipose
* No acceptance of study

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients of ambulatory of Sleep Respiratory Disorders of Santa Casa de Limeira
Sampling Method: Probability Sample
Enrollment: 159 (Actual)
Dates: Start 2007-01; Primary Completion 2008-02 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Stanford Classification for snoring | One year

SECONDARY OUTCOMES:
Apnea-Hyponea Index | one year

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Dia, Limeira, S, Brazil